CLINICAL TRIAL: NCT06314724
Title: Immunogenicity and Safety of Varicella Vaccine, Live in Healthy Children Aged 12~15 Months in the Philippines: a Randomized, Double-blind, Active-controlled Phase Ⅲ Clinical Trial
Brief Title: Immunogenicity and Safety of Varicella Vaccine, Live in Healthy Children Aged 12~15 Months in the Philippines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sinovac (Dalian) Vaccine Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO-VZV-4006
Record Dates: First submitted 2024-03-06; First posted 2024-03-18 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Varicella
MeSH Terms: conditions — Chickenpox | interventions — Chickenpox Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Varicella vaccine group (Experimental): Participants will receive a single dose of investigational varicella vaccine on Day 0.
  Interventions: Biological: Varicella Vaccine
- Varivax (Active Comparator): Participants will receive a single dose of Varivax on Day 0.
  Interventions: Biological: Varivax

INTERVENTIONS:
Biological: Varicella Vaccine — lyophilized powder,subcutaneous injection
  Arms: Varicella vaccine group
Biological: Varivax — lyophilized powder,subcutaneous injection
  Arms: Varivax

SUMMARY:
This is a Phase Ⅲ, randomized, double-blind, active-controlled study to assess the immunogenicity and safety of the varicella vaccine,Live (hereinafter referred to as "varicella vaccine")manufactured by Sinovac (Dalian) Vaccine Technology Co., LTD.(hereinafter referred to as "Sinovac").

DETAILED DESCRIPTION:
A total of 642 healthy participants aged 12~15 months will be enrolled. All participants will be randomized at a 1:1 ratio to receive a single dose of varicella vaccine either manufactured by Sinovac (Group A) or Merck Sharp & Dohme (MSD, Group B).

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 12~15 months;
* Participants' legal guardians are able to understand and sign the informed consent voluntarily;
* Participants are able to comply with the study procedures based on the assessment of the investigator;
* Participants should provide verifiable identification, to be contacted, and to contact the investigator during the study period.

Exclusion Criteria:

* Prior vaccination with any varicella containing vaccines;
* Prior history of VZV infection;
* Known allergy to vaccines or vaccine ingredients, or serious adverse reactions to vaccines, such as urticaria, dyspnea, angioneurotic edema;
* Autoimmune diseases (including but not limited to systemic lupus erythematosus, rheumatoid arthritis, etc.) or immunodeficiency/immunosuppression (such as HIV infection, organ transplantation), asplenia;
* Receipt of blood products or immunoglobulins within the past 3 months before enrollment in this study, or scheduled to receive these treatments during the study period;
* Receipt of other investigational vaccines within 30 days prior to vaccination in this study;
* Receipt of attenuated live vaccines within 28 days prior to vaccination in this study;
* Receipt of inactivated or subunit vaccines within 7 days prior to vaccination in this study;
* Acute onset of various acute diseases or chronic diseases within 7 days prior to vaccination in this study;
* Has fever on the day of vaccination, with the axillary temperature >37°C before vaccination;
* Is participating in or planning to participate in other vaccine or drug clinical trials;
* Any confirmed or suspected syphilis, hepatitis B or hepatitis C infection;
* According to the investigator's judgment, the subject has any other factors that might interfere with the clinical trial results or pose additional risk to the participant due to participation in the study.

Ages: 12 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 642 (Actual)
Dates: Start 2024-02-29 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-09-06 (Actual)

PRIMARY OUTCOMES:
Seroresponse rate of varicella-zoster virus (VZV) antibody | Day 42 after vaccination
  The seroresponse rate of VZV antibodies on Day 42 after vaccination among susceptible population.

SECONDARY OUTCOMES:
Geometric mean concentrations (GMCs) of VZV antibody | Day 42 after vaccination after vaccination
  The GMC of VZV antibodies on Day 42 after vaccination among susceptible population.
GMC of VZV antibody | Day 42 after vaccination
  The GMC of VZV antibodies on Day 42 after vaccination among among all participants.
seropositive rate | Day 42 after vaccination
  The seropositive rate of VZV antibodies on Day 42 after vaccination among all participants.
Geometric mean fold rise (GMFR) from before vaccination of VZV antibody | Day 42 after vaccination
  The GMFR from before vaccination of VZV antibodies on Day 42 after vaccination among all participants.
Incidence of adverse reactions within 0~42 days after vaccination | Within 0~42 days after vaccination
  Incidence of adverse reactions within 0~42 days after vaccination among all participants
Incidence of adverse reactions within 0~14 days after vaccination | Within 0~14 days after vaccination
  Incidence of adverse reactions within 0~14 days after vaccination among all participants
Incidence of serious adverse events (SAE) within 0~42 days after vaccination | Within 0~42 days after vaccination
  Incidence of SAE within 0~42 days after vaccination among all participants.

CONTACTS AND LOCATIONS:
Overall Officials: Rommel Crisenio M. Lobo, MD, Principal Investigator — Cardinal Santos Medical Center; Nancy Nazaire Bermal, MD, Principal Investigator — San Juan de Dios Educational Foundation, lnc.-Hospital
Locations (2):
- Philippines (2):
  - San Juan de Dios Educational Foundation, lnc., Pasay
  - Cardinal Santos Medical Center, San Juan City